CLINICAL TRIAL: NCT00904306
Title: Chromium Picolinate in Binge Eating Disorder: A Feasibility Study
Brief Title: Binge Eating and Chromium Study
Acronym: BEACh
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Kimberly Brownley, Assistant Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3062-04003; 08-0953 (GCRC #2713)
Record Dates: First submitted 2009-05-17; First posted 2009-05-19 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Binge Eating Disorder
Keywords: binge eating; chromium; mood; glucose; appetite
MeSH Terms: conditions — Binge-Eating Disorder; Bulimia | interventions — Sugars; picolinic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sugar pill (Placebo Comparator): 6 months treatment with placebo
  Interventions: Dietary Supplement: Sugar Pill
- low dose (Active Comparator): 600ug/day chromium picolinate for 6 months
  Interventions: Dietary Supplement: chromium picolinate
- high dose chromium picolinate (Active Comparator): 1000 ug/day
  Interventions: Dietary Supplement: chromium picolinate

INTERVENTIONS:
Dietary Supplement: Sugar Pill — placebo oral tablet taken once per day
  Arms: Sugar pill
Dietary Supplement: chromium picolinate — 1000 ug/day chromium picolinate for 6 months
  Arms: high dose chromium picolinate
Dietary Supplement: chromium picolinate — 600 ug/day chromium picolinate
  Arms: low dose

SUMMARY:
The purpose of this study is to test the feasibility and preliminary efficacy of a 6-month chromium picolinate (CrPic) treatment trial in binge eating disorder (BED).

DETAILED DESCRIPTION:
Binge eating (i.e., the consumption of unusually large amounts of food with a sense of loss of control) is a common problem with serious public health implications in large part due to its role in obesity. Binge eating leads to weight gain and is common in overweight individuals. Current treatments for binge eating disorder (BED) are inadequate, and previous randomized treatment trials have suffered from high drop out rate due to the adverse effects of pharmacological agents. Chromium picolinate is a dietary supplement that has been shown to reduce symptoms of depression and appetite regulation problems in patients with atypical depression; chromium picolinate also affects insulin regulation and has been shown to improve glucose levels in patients with type-2 diabetes. This pilot study will evaluate the effect of chromium picolinate on binge eating, mood, body weight, and glucose regulation in overweight individuals with BED.

ELIGIBILITY:
Inclusion Criteria:

1. Currently meets DSM-IV criteria for binge eating disorder (BED);
2. Is able to provide informed consent and meet study visit requirements; and
3. Is psychiatrically stable (e.g., no current suicidal or homicidal intent or other psychiatric condition that requires acute intervention).

Exclusion Criteria:

1. Body mass index (BMI) < 24.9 kg/m^2 (underweight or normal weight) or ≥ 40 kg/m^2 (severely obese);
2. Postmenopausal;
3. Age < 18 or > 55 years;
4. Pregnant, planning on becoming pregnant during the study period, or lactating;
5. Current psychotropic medication use;
6. Current use of insulin or other medications to control glucose metabolism;
7. Current use of medications known to significantly influence appetite or weight [i.e., over-the-counter appetite suppressants that contain phentermine or sibutramine, atypical antipsychotic agents with high weight gain liability (such as olanzapine, risperidone, etc), prednisone, etc.];
8. Fasting glucose level > 126 mg/dL (indicative of diabetes); and
9. Creatinine level indicating renal insufficiency (> 1.0 for women; > 1.2 for men).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2008-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
binge eating frequency | baseline, 3 and 6 months, 3-month followup

SECONDARY OUTCOMES:
mood | baseline, 3 adn 6 months, 3-month followup
insulin sensitivity | baseline, 3 adn 6 months, 3-month followup
body weight | baseline, 3 adn 6 months, 3-month followup

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Brownley, PhD, Principal Investigator — University of North Carolina, Chapel Hill

REFERENCES:
- [Background] Brownley KA, Berkman ND, Sedway JA, Lohr KN, Bulik CM. Binge eating disorder treatment: a systematic review of randomized controlled trials. Int J Eat Disord. 2007 May;40(4):337-48. doi: 10.1002/eat.20370. PMID 17370289
- [Background] Bulik CM, Brownley KA, Shapiro JR. Diagnosis and management of binge eating disorder. World Psychiatry. 2007 Oct;6(3):142-8. PMID 18188431
- [Background] Berkman ND, Bulik CM, Brownley KA, Lohr KN, Sedway JA, Rooks A, Gartlehner G. Management of eating disorders. Evid Rep Technol Assess (Full Rep). 2006 Apr;(135):1-166. PMID 17628126
- [Derived] Brownley KA, Von Holle A, Hamer RM, La Via M, Bulik CM. A double-blind, randomized pilot trial of chromium picolinate for binge eating disorder: results of the Binge Eating and Chromium (BEACh) study. J Psychosom Res. 2013 Jul;75(1):36-42. doi: 10.1016/j.jpsychores.2013.03.092. Epub 2013 Apr 22. PMID 23751236